CLINICAL TRIAL: NCT00820872
Title: Phase II Safety Study of Docetaxel and Carboplatin in Combination With Trastuzumab and Lapatinib in Early Breast Cancer
Brief Title: Docetaxel, Carboplatin, Trastuzumab, and Lapatinib in Treating Patients With Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N083E; NCI-2009-00671 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000631625 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Carboplatin; Docetaxel; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + carboplatin + trastuzumab + lapatinib (Experimental): Patients receive docetaxel IV over 60 minutes and carboplatin IV over 30 minutes on day 1, trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15, and oral lapatinib ditosylate on days 1-21 (TCHL). Treatment with TCHL repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30-90 minutes on day 1 and oral lapatinib ditosylate on days 1-21 (days 1-7 of course 12 only) (LT). Treatment with LT repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 8 years.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: docetaxel; Drug: lapatinib ditosylate

INTERVENTIONS:
Biological: trastuzumab
Drug: carboplatin
Drug: docetaxel
Drug: lapatinib ditosylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel together with carboplatin, trastuzumab, and lapatinib may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving docetaxel together with carboplatin, trastuzumab, and lapatinib in treating patients with early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability (including the rate of diarrhea) of adjuvant therapy comprising docetaxel, carboplatin, trastuzumab (Herceptin®), and lapatinib ditosylate in patients with early-stage breast cancer.

Secondary

* Evaluate the adverse event profile of this regimen in these patients.
* Evaluate LVEF in patients receiving this regimen.

OUTLINE: Patients receive docetaxel IV over 60 minutes and carboplatin IV over 30 minutes on day 1, trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15, and oral lapatinib ditosylate on days 1-21 (TCHL). Treatment with TCHL repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30-90 minutes on day 1 and oral lapatinib ditosylate on days 1-21 (days 1-7 of course 12 only) (LT). Treatment with LT repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity..

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive adenocarcinoma of the breast fulfilling the following criteria:

  * Nonmetastatic disease
  * Operable and adequately excised

    * Patients with nonresectable deep margin invasion are eligible provided they have had or will receive radiotherapy to the region
    * Patients with histologically documented infiltration of the skin (pT4) are eligible provided they have undergone or will receive radiotherapy encompassing the tumor bed
  * Node-positive OR -negative and determined eligible to receive adjuvant trastuzumab (Herceptin®)
* No positive or suspicious internal mammary nodes by SNS that have not been or will not be irradiated
* No supraclavicular lymph node involvement (confirmed by fine needle aspiration or biopsy)
* Over expression and/or amplification of HER2 in the invasive component of the primary tumor, according to one of the following:

  * 3+ over-expression by IHC (> 30% of invasive tumor cells)
  * 2+ or 3+ (in 30% or less neoplastic cells) over-expression by IHC AND in situ hybridization (FISH/CISH) test demonstrating HER2 gene amplification
  * HER2 gene amplification by FISH/CISH (> 6 HER2 gene copies per nucleus, or a FISH ratio [HER2 gene copies to chromosome 17 signals] of > 2.2.)

    * Negative or equivocal overall result (FISH test ratio of < 2.2, < 6.0 HER2-gene copies per nucleus) and staining scores of 0, 1+, 2+, or 3+ (in 30% or less neoplastic cells) by IHC not allowed
* Hormone receptor status known (estrogen receptor with or without progesterone receptor)

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-1
* Hemoglobin ≥ 10.0 g/dL
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN (≤ 2.0 times ULN if known Gilbert syndrome)
* Baseline LVEF ≥ 50% measured by ECHO or MUGA scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious cardiac illness or medical condition including, but not limited to, any of the following:

  * History of documented congestive heart failure (any NYHA class) or systolic dysfunction (LVEF < 50%)
  * High-risk uncontrolled arrhythmias (e.g., ventricular tachycardia, high-grade atrioventricular-block [second degree or higher], or supraventricular arrhythmias that are not adequately rate-controlled)
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly controlled hypertension (any reading of systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg)
* No other concurrent serious diseases that may interfere with planned treatment including severe pulmonary conditions or illness
* None of the following:

  * Ulcerative colitis
  * Malabsorption syndrome
  * Any disease significantly affecting gastrointestinal function
  * Inability to swallow oral medication

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior mediastinal irradiation except internal mammary-node irradiation for the present breast cancer
* No prior anti-HER2 therapy for any reason
* No prior biologic or immunotherapy for breast cancer
* No prior resection of the stomach or small bowel
* No other concurrent anticancer therapy including chemotherapeutic agents, biologic agents, or radiotherapy
* No concurrent anticancer treatment in another investigational trial with hormone therapy or immunotherapy unless approved by the study chair
* No concurrent CYP3A4 inhibitors or inducers
* No concurrent epoetin alfa, including darbepoetin alfa
* No concurrent oprelvekin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (136):
- United States (136):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Patients receive docetaxel IV over 60 minutes and carboplatin IV over 30 minutes on day 1, trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15, and oral lapatinib ditosylate on days 1-21 (TCHL). Treatment with TCHL repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30-90 minutes on day 1 and oral lapatinib ditosylate on days 1-21 (days 1-7 of course 12 only) (LT). Treatment with LT repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 8 years.
Period: Overall Study
Arm/Group | Group 1
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: Years] | 54.5 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing Grade 3 or 4 Diarrhea as Measured by NCI CTCAE v3.0
Time Frame: Up to 10 years
Population: All evaulable patients
Measure: Number; unit: percentage of patients
Arm/Group | Group 1
Number analyzed (Participants) | 30
percentage of patients | 43

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=30)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=30)
Hemoglobin decreased (Blood and lymphatic system disorders) | 27 (219)
Hemolysis (Blood and lymphatic system disorders) | 1 (3)
Left ventricular dysfunction (Cardiac disorders) | 3 (8)
Left ventricular failure (Cardiac disorders) | 3 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 28 (180)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 14 (47)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (4)
Mucositis oral (Gastrointestinal disorders) | 10 (30)
Nausea (Gastrointestinal disorders) | 24 (104)
Vomiting (Gastrointestinal disorders) | 19 (38)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 25 (195)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 4 (11)
Opportunistic infection (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 16 (47)
Alkaline phosphatase increased (Investigations) | 13 (58)
Aspartate aminotransferase increased (Investigations) | 12 (40)
Bilirubin increased (Investigations) | 5 (23)
Coagulopathy (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 3 (10)
Lymphocyte count decreased (Investigations) | 2 (13)
Neutrophil count decreased (Investigations) | 17 (74)
Platelet count decreased (Investigations) | 19 (76)
Weight gain (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (29)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (63)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (99)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (15)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (15)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (5)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 15 (68)
Hot flashes (Vascular disorders) | 1 (2)
Lymphedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes